CLINICAL TRIAL: NCT04725019
Title: Enhancing Motor Learning in Children With Cerebral Palsy Using Transcranial Direct-current Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Claudio, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5825
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + motor training (Experimental): In this arm, participants will receive 20 minutes of active tDCS and motor training that involves a high number of repetitions while engaged in child-friendly games.
  Interventions: Device: active transcranial direct current stimulation; Behavioral: Motor training
- Sham tDCS + motor training (Experimental): In this arm, participants will receive 20 minutes of sham tDCS and motor training that involves a high number of repetitions while engaged in child-friendly games. Children receiving sham tDCS will wear the tDCS device but not receive active stimulation.
  Interventions: Behavioral: Motor training

INTERVENTIONS:
Device: active transcranial direct current stimulation — Participants will receive 20 min of tDCS over the scalp during 20 min of motor training.
  Arms: Active tDCS + motor training
Behavioral: Motor training — Participants will engage in a high number of repetition of movements that use both hands while playing with toys and games. Training will be provided 20 min/day, for 5 consecutive days.

SUMMARY:
The goal of this study is to test the effects of transcranial direct current stimulation (tDCS) on motor learning and brain plasticity in children with unilateral spastic cerebral palsy (USCP).

ELIGIBILITY:
Inclusion Criteria:

Children between 6-17 years old who have been diagnosed with cerebral palsy, with the following joint mobility: wrist extension 20º, metacarpophalangeal and proximal interphalangeal joints 10º. Ability to cooperate and follow simple directions.

Exclusion Criteria:

* Seizure beyond age 2, use of anti-seizure medication, history or family history of epilepsy, cranial metal implants, structural brain lesion, devices that may be affected by tDCS or TMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* True positive response on the Transcranial Magnetic Stimulation and MRI Safety Screen
* Current use of medications known to lower the seizure threshold
* Previous episode of unprovoked neurocardiogenic syncope
* Indwelling metal or incompatible medical devices
* Centrally-acting medications including anti-seizure medications
* Evidence of scalp disease or skin abnormalities
* Current medical illness unrelated to CP
* High motor ability in affected arm (i.e. no asymmetry in scores of hand function)
* Severe spasticity
* Lack of asymmetry in hand function
* Orthopedic surgery in affected arm
* Botulinum toxin therapy in either upper extremity during last 6 months, or planned during study period
* Currently receiving intrathecal baclofen
* History of broken arm (either arm) 1 year prior to study enrollment

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Assisting Hand Assessment | Day before intervention begins, compared to day after intervention ends (approximately 1 week)
  Investigators will measure changes in how well the child uses both hands cooperatively for bimanual activities.
Changes in the Box and Blocks test | Day before intervention begins, compared to day after intervention ends (approximately 1 week)
  Investigators will measure changes in the movement speed of the hands.

SECONDARY OUTCOMES:
Changes in Motor-evoked Potential assessment | Day before intervention begins, compared to day after intervention ends (approximately 1 week)
  Investigators will measure change in measurements of cortical excitability using transcranial magnetic stimulation (TMS) from baseline to follow-up (1 week).

IPD SHARING:
Plan to Share IPD: Undecided
If the study is funded by National Institute of Health (NIH), the investigators will share individual participant data (IPD) via the NIH Data Hub (DASH), which is sponsored by the National Institute of Child Health and Development (NICHD).